CLINICAL TRIAL: NCT05070065
Title: VIVA-CORE! Virtual Reality VAlidation Tool for Cognitive Rehabilitation, a REcovery Oriented Project for People With Psychosocial Disabilieties: Protocol of Randomize Clinical Trial
Brief Title: Virtual Reality VAlidation Tool for Cognitive Rehabilitation, Oriented Project for People With Psychosocial Disabilieties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Mauro Giovanni Carta, Professor, University of Cagliari
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Prot. PG/2020/7577
Record Dates: First submitted 2021-07-21; First posted 2021-10-06 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Mood Disorders
Keywords: Virtual Reality; Remediation; Mental Health; Recovery
MeSH Terms: conditions — Mood Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized controlled open-label cross-over clinical feasibility study with waiting list
Who Masked: Participant
Masking Description: people with psychosocial disabilities
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): The experimental group A receives the cognitive remedy intervention with virtual reality (CEREBRUM)
  Interventions: Device: Cognitive remedy intervention with virtual reality (CEREBRUM)
- waiting list (Other): waiting list
  Interventions: Device: Cognitive remedy intervention with virtual reality (CEREBRUM)

INTERVENTIONS:
Device: Cognitive remedy intervention with virtual reality (CEREBRUM) — Cognitive Remedial method Virtual Reality (CEREBRUM)

SUMMARY:
Randomized controlled open-label cross-over clinical feasibility study with waiting list, 60 people will be recruited from the Consultation and Psychosomatic Psychiatry Center of the University Hospital of Cagliari (San Giovanni di Dio Civil Hospital) with a diagnosis of mental disorder. The investigators propose a VR intervention of 3 months with 2 weekly session of CEREBRUM (cognitive remedy intervention with virtual reality) first to the group A and then to the group B.

DETAILED DESCRIPTION:
Background: Cognitive remedial interventions have been found to be effective in the treatment of various psycho-social disorders. The use of Virtual reality as a rehabilitation tool has been showing various scientific evidences in recent years like in cardiovascular, neurological and musculoskeletal rehabilitation. In mental health evidence they seem to be concentrated in the rehabilitation of social cognition in people with schizophrenia diagnosis and psychotherapy. The aim of this study is to evaluate the feasibility and the effectiveness of the first Cognitive Remedial toll in Virtual Reality (CEREBRUM) for people that has experienced in mental health.

Methods: Randomized controlled open-label cross-over clinical feasibility study with waiting list, 60 people will be recruited from the Consultation and Psychosomatic Psychiatry Center of the University Hospital of Cagliari (San Giovanni di Dio Civil Hospital) with a diagnosis of mental disorder. The investigators propose a intervention of 3 months with 2 weekly session of CEREBRUM first to the group A and then to the group B

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75;
* Diagnosis of psychosis and / or mood disorder according to DSM-IV (American Psychiatric Association, 2000).
* both sexes;
* users who sign the informed consent;
* users under protection for which the informed consent is signed by the guardian

Exclusion Criteria:

* The non-satisfaction of the inclusion criteria;
* The diagnosis of epilepsy or serious eye diseases, due to the risk associated with the excessive stimulation of virtual reality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Memory | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Rey's Figure Test Word's Figure Test Digit Span Forward and Backward Test Test of the Tale
Monitoring Side effects of Virtual Reality | During the first VR session - At 1 month (after 8 sessions) - T1 (at 3 months from baseline)
  Questionnaire (Qualitative)
Attention | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Matrix Test Digit Symbol Substitution Test
Executive functions | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Trial Making Test Verbal Phonological and Semantic Fluency Test Cognitive Estimation Test - CET Stroop Test Frontal Assessment Battery - FAB

SECONDARY OUTCOMES:
Quality of Life | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Short Form Healthy Survey Questionnaire - SF-12
Alexithymia | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Toronto Alexithymia Scale - TAS-20
Anxiety | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Self Anxiety Rating Scale - SAS
Depression | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  The Patient Health Questionnaire - PHQ-9
Biological Rythms | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Biological Rythms Interview of Assesment in Neuropsychiatry - BRIAN
General and social functioning | All measure at: T0 (base line) -T1 (at 3 months from baseline) -T2 (at 6 months from baseline) -T3 (at 12 months from baseline)
  Health of the Nation Outcome Scales - HoNOS

CONTACTS AND LOCATIONS:
Locations (1):
- P.O. San Giovanni di Dio, AOU Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sancassiani F, Perra A, Galetti A, Di Natale L, De Lorenzo V, Lorrai S, Kalcev G, Pintus E, Cantone E, Nonnis M, Nardi AE, Montisci R, Primavera D. Alexithymia and Bipolar Disorder: Virtual Reality Could Be a Useful Tool for the Treatment and Prevention of These Conditions in People with a Physical Comorbidity. J Clin Med. 2024 Oct 18;13(20):6206. doi: 10.3390/jcm13206206. PMID 39458156
- [Derived] Perra A, De Lorenzo V, Zaccheddu R, Locci A, Piludu F, Preti A, Di Natale L, Galetti A, Nardi AE, Cossu G, Sancassiani F, Barbato S, Cesaretti O, Kurotshka PK, Carta MG. Cognitive Remediation Virtual Reality Tool a Recovery-Oriented Project for People with Bipolar Disorder: Protocol of a Feasibility Randomized Clinical Trial. Clin Pract Epidemiol Ment Health. 2022 Oct 6;18:e174501792208220. doi: 10.2174/17450179-v18-e2208220. eCollection 2022. PMID 37274852
- [Derived] Perra A, Galetti A, Zaccheddu R, Locci A, Piludu F, Preti A, Primavera D, Di Natale L, Nardi AE, Kurotshka PK, Cossu G, Sancassiani F, Stella G, De Lorenzo V, Zreik T, Carta MG. A Recovery-Oriented Program for People with Bipolar Disorder through Virtual Reality-Based Cognitive Remediation: Results of a Feasibility Randomized Clinical Trial. J Clin Med. 2023 Mar 9;12(6):2142. doi: 10.3390/jcm12062142. PMID 36983145